CLINICAL TRIAL: NCT06633965
Title: Safety and Feasibility Testing of a Smaller Network Version of AIDANET (MiniNET)
Brief Title: Safety and Feasibility Testing of a Smaller Network Version of AIDANET
Acronym: MiniNET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marc Breton (Other)
Collaborators: Tandem Diabetes Care, Inc. (Industry); DexCom, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Marc Breton, Professor, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 301828
Record Dates: First submitted 2024-10-04; First posted 2024-10-09 (Actual); Results first posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Meal Boluses; Fully Closed Loop (FCL); AIDANET
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to assess a 1-week usual care period before use of the AIDANET system (Group A) or after use of the AIDANET system (Group B).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Usual Care→AIDANET (Active Comparator): Participants will complete 7 days/6 nights at home usual care period using their personal equipment. Participants will then use the AIDANET system during a 3 days/2 nights hotel admission. Participants will continue to use the AIDANET system at home for 7 days/6 nights.
  Interventions: Device: AIDANET
- AIDANET→Usual Care (Active Comparator): Participants will use AIDANET system during a 3 days/2 nights hotel admission. Participants will continue to use the AIDANET system at home for 7 days/6 nights and then will complete 7 days/6 nights at home usual care period using their personal equipment.
  Interventions: Device: AIDANET

INTERVENTIONS:
Device: AIDANET — AIDANET is a fully automated, utilizing a Bolus Priming System (BPS) that recognizes meal ingestion and delivers a quick priming dose of insulin prior to extreme blood sugar excursions.
  Other Names: Group B
  Arms: AIDANET→Usual Care
Device: AIDANET — AIDANET is a fully automated, utilizing a Bolus Priming System (BPS) that recognizes meal ingestion and delivers a quick priming dose of insulin prior to extreme blood sugar excursions.
  Other Names: Group A
  Arms: Usual Care→AIDANET

SUMMARY:
A randomized 1:1 crossover trial that intends to demonstrate feasibility and safety of the Automated Insulin Delivery as Adaptive NETwork (AIDANET) system run in a new smaller network version, used in full closed loop (FCL) by adults who have been diagnosed with type 1 diabetes (T1D).

DETAILED DESCRIPTION:
The study will be performed for about 36 hours at a local hotel. Following the hotel session, participants will undergo a 7 day/6-night Remote Monitored At-Home use session. A one-week control period gathering data on glycemic control and insulin administration with the participants usual care therapy will also be completed. Participants will be randomized 1:1, to either Group A (control period prior to AIDANET use) or Group B (control period after AIDANET use).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18.0 and ≤60 years old at time of consent
2. Clinical diagnosis, based on investigator assessment, of type 1 diabetes for at least one year
3. Currently using insulin pump for at least three months; Any pump, either open loop or hybrid closed loop may be used.
4. Currently using insulin for at least six months.
5. Willingness to switch to use a commercially approved personal insulin (e.g., lispro or aspart, or biosimilar approved products) within the study pump as directed by the study team.
6. Currently using a Dexcom G6 or G7 CGM.
7. Has one or more supportive companions knowledgeable about emergency procedures for severe hypoglycemia and able to contact emergency services and study staff that either lives with participant or located within approximately 30 minutes of participant and able to locate participant in the event of an emergency.
8. Participant not currently known to be pregnant or breastfeeding.
9. If participant capable of becoming pregnant, must agree to use a form of contraception to prevent pregnancy while a participant in the study (e.g. hormonal contraception, abstinence from heterosexual intercourse). A negative serum or urine pregnancy test will be required for all females of childbearing potential. Participants who become pregnant will be discontinued from the study. Also, participants who during the study develop and express the intention to become pregnant within the timespan of the study will be discontinued.
10. Willingness to use the study FCL system (CGM, pump, and phone) during the relevant study period.
11. Willingness not to start any new non-insulin glucose-lowering agent during the course of the trial.
12. Willingness to participate in all study procedures including the house/hotel session, exercise challenges (e.g., one hour per day during hotel), and to consume approximately 3 unannounced meals per day during the relevant portion of the supervised hotel session.
13. Access to internet at home and willingness to upload data during the study as needed.
14. Investigator has confidence that the participant can successfully operate all study devices and is capable of adhering to the protocol.
15. Participant is proficient in reading and writing English.

Exclusion Criteria:

1. Plans to start a new non-insulin glucose-lowering agent (e.g., GLP-1 receptor agonists, Symlin, DPP-4 inhibitors, sulfonylureas). Participants may be on a stable dose of such an agent for at least the past month.
2. Current use of an SGLT-2 or SGLT-1/2 inhibitor due to risk of euglycemic DKA.
3. Hemophilia or any other bleeding disorder.
4. History of severe hypoglycemic events with seizure or loss of consciousness in the last 12 months.
5. History of DKA event in the last 12 months.
6. History of chronic renal disease (Stage 4 or unstable Stage 3b per investigator judgment) or currently on peritoneal or hemodialysis.
7. History of adrenal insufficiency.
8. Currently being treated for a seizure disorder.
9. Hypothyroidism or hyperthyroidism that is not adequately treated.
10. Coronary artery disease or other heart condition that would prevent participation in moderate intensity exercise.
11. Use of oral or injectable steroids at the time of enrollment or within the last 4 weeks.
12. Planned surgery during the study period.
13. Known ongoing adhesive intolerance that is not well managed.
14. A condition, which in the opinion of the investigator or designee, would put the participant or study at risk.
15. Participation in another interventional trial at the time of enrollment.
16. Participant with a direct supervisor involved in the conduct of the trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2024-11-20 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2024-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sue Brown, MD, Principal Investigator — University of Virginia Center for Diabetes Technology
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Will follow the NIH Data Sharing Policy and Implementation Guidance on sharing research resources for research purposes to qualified individuals in the scientific community.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available after the publication of the manuscript.
Access Criteria: The Data Sharing Agreements will be formulated by the study team

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eight participants with T1D provided informed consent. One did not pass the screening process and another withdrew prior to the study intervention. The remaining six participants were randomized and completed the trial in December 2024.
Period: Overall Study
Arm/Group | Usual Care→AIDANET | AIDANET→Usual Care
Started | 4 | 3
Completed | 4 | 2 (One subject withdrew before study intervention)
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: One subject withdrew prior to study intervention. Results were only analyzed for subjects who started data collection.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care→AIDANET | AIDANET→Usual Care | Total
Number analyzed (Participants) | 4 | 2 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 6
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (6.5) | 36.5 (8.5) | 40.3 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 2 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 2 | 6
Percentage of HbA1c (%) [Mean (Standard Deviation); unit: percentage] | 7.1 (0.5) | 7.3 (0.1) | 7.17 (0.41)
Weight (kg) [Mean (Standard Deviation); unit: kilograms] | 81.3 (17.5) | 87.5 (0.5) | 83.4 (14.6)
BMI (kg/m2) [Mean (Standard Deviation); unit: kilograms per square-meter] | 27.7 (3.0) | 33.8 (1.5) | 29.7 (3.9)
Diabetes duration (y) [Mean (Standard Deviation); unit: years] | 21.6 (8.2) | 31.4 (5.3) | 24.9 (8.7)
CGM use [Count of Participants; unit: Participants]
  Dexcom G6 | 2 | 1 | 3
  Dexcom G7 | 2 | 1 | 3
Pump use [Count of Participants; unit: Participants]
  Tandem /t:slim X2 with Control IQ | 2 | 2 | 4
  Insulet / Omnipod 5 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in the Mean Continuous Glucose Monitor (CGM) Between the Week of the Usual Care Observational Period and the Week of AIDANET At-Home.
Description: This study represents a small pilot study to assess the safety and efficacy of the small-version AIDANET system and is not formally powered. Nevertheless, the randomized crossover design will allow for analysis of period effects between Group A and Group B. Comparison between these groups will be made to determine if a period effect can explain part of the benefit of the FCL system during the at-home period.
Time Frame: 2 weeks
Population: One participant withdrew prior to study intervention. Results were only analyzed for participants who started and completed data collection.
Measure: Mean (Standard Deviation); unit: miligrams per deciliter
Arm/Group | Usual Care→AIDANET | AIDANET→Usual Care
Number analyzed (Participants) | 4 | 2
miligrams per deciliter | -6.8 (15.1) | -2.1 (20.7)

2. Secondary Outcome: Difference in Percent Time-in-range
Description: Difference in percent CGM samples in 70-180 mg/dL between the Week of the Usual Care Observational Period and the Week of AIDANET At-home. Represented as AIDANET minus Usual Care.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: percentage of time-in-range
Arm/Group | Usual Care→AIDANET | AIDANET→Usual Care
Number analyzed (Participants) | 4 | 2
percentage of time-in-range | 1.55 (4.34) | 2.76 (10.6)

3. Secondary Outcome: Difference in Percent Time-below-range
Description: Difference in CGM percent samples < 70mg/dL between the Week of the Usual Care Observational Period and the Week of AIDANET At-home. Represented as AIDANET minus Usual Care.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: percentage of time-below-range
Arm/Group | Usual Care→AIDANET | AIDANET→Usual Care
Number analyzed (Participants) | 4 | 2
percentage of time-below-range | 0.93 (2.10) | 0.06 (0.45)

4. Secondary Outcome: Difference in Percent Time-in-tight-range
Description: Difference in percent CGM samples in 70-140 mg/dL between the Week of the Usual Care Observational Period and the Week of AIDANET At-home. Represented as AIDANET minus Usual Care.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: percentage of time-in-tight-range
Arm/Group | Usual Care→AIDANET | AIDANET→Usual Care
Number analyzed (Participants) | 4 | 2
percentage of time-in-tight-range | 1.69 (10.71) | 4.01 (7.19)

ADVERSE EVENTS:
Time Frame: 24 days. Three days of hotel use with AIDANET followed by 7 days of AIDANET use at home, and 14 days of Usual Care
Arm/Group | Usual Care→AIDANET | AIDANET→Usual Care
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/2
Other Adverse Events (participants affected / at risk) | 0/4 | 0/2

LIMITATIONS AND CAVEATS:
This study represents a small pilot study to assess the safety and efficacy of the small-version AIDANET system and is not formally powered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-10-25): https://cdn.clinicaltrials.gov/large-docs/65/NCT06633965/Prot_SAP_001.pdf
  • Informed Consent Form (2024-11-12): https://cdn.clinicaltrials.gov/large-docs/65/NCT06633965/ICF_000.pdf